CLINICAL TRIAL: NCT05354752
Title: Randomized, Double-blind, Multiple-dose Escalation, Placebo-controlled Phase I Clinical Study to Evaluate the Tolerance, Pharmacokinetics and Pharmacodynamics of VC005 Tablets in Healthy Subjects
Brief Title: Multiple-dose Escalation Clinical Study of VC005 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-102
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: healthy subjects
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VC005 Tablets Dose escalation groups (Experimental): VC005 Tablets groups Repeat doses
  Interventions: Drug: VC005 tablets
- VC005 Tablets Placebo groups (Placebo Comparator): VC005 Tablets Placebo groups Repeat doses.
  Interventions: Drug: VC005 Placebo tablets

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 7 days
  Arms: VC005 Tablets Dose escalation groups
Drug: VC005 Placebo tablets — VC005 placebo groups repeat administration for 7 days
  Arms: VC005 Tablets Placebo groups

SUMMARY:
This clinical trial is a randomized, double-blind, single-center, placebo-controlled and multiple-dose escalation Pharmacokinetics study

DETAILED DESCRIPTION:
The main purpose of this trial is to evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of VC005 Tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 to 45 years old，inclusive
2. Male subjects weighing at least 50 kg and female subjects weighing at least 45 kg. Body mass index (BMI) between 18 and 28 kg/m2, inclusive
3. During the trial and within 3 months after the completion of the trial (the time should exceed the time required for sperm production), there is no fertility plan, and is willing to use effective contraceptive measures (non hormonal contraceptive measures) and there is no sperm donation and egg donation plan
4. Volunteer to participate in the trial and sign an informed consent form
5. Subjects who are able to communicate well with the investigator are willing and able to comply with all planned visits, treatment plans, laboratory examinations and other research procedures
6. Physical examination and vital signs are normal or abnormal with no clinical significance

Exclusion Criteria:

1. Suspected to be allergic to the study drug or any component in the study drug, or allergic constitution
2. abnormal electrocardiogram with clinical significance
3. Those who have evidence of atypical hyperplasia or a history of malignant tumor
4. Suffer from eye diseases, including history of eye surgery or laser surgery (except laser surgery for myopia)
5. Those who have a history of herpes simplex or herpes zoster 3 months before administration
6. Have any history or evidence of active tuberculosis (TB) or latent TB infection (TB enzyme-linked immunospot test (T-SPOT. TB) positive), or have a history of previous skin TB test or QuantiFERON TB gold in tube test (GIT analysis) positive
7. Known active bacteria, viruses, fungi, parasitic infections or other infections or any infections that require antibiotic treatment or hospitalization (4 weeks before screening), or any acute infections within 2 weeks of baseline
8. Those who have participated in clinical trials of any drug or medical device (including the placebo group) within 3 months before screening
9. Those who have been vaccinated within 2 weeks before administration, or plan to be vaccinated during the study period
10. Those who are usually anorexia, dieting, or have started a significantly abnormal diet (such as dieting) within 4 weeks before screening; those who cannot follow a uniform diet or have difficulty swallowing
11. Those who have undergone any surgeries within 6 months before screening
12. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines within 14 days before screening
13. Those who use any drug that inhibits or induces liver enzyme activity within 28 days before administration or during the study period
14. Those who were in blood donation within 3 months before screening and donated blood volume ≥400 mL, or received blood transfusion
15. Those who with dyslipidemia of clinical significance and coronary heart disease
16. Pregnant and lactating females, or females who have a positive pregnancy test
17. Those who have difficulty in blood collection or cannot tolerate venipuncture, and those who have a history of fainting needles and bleeding
18. Those who smoke ≥ 5 cigarettes per day within 3 months before screening and cannot stop using any tobacco products from the end of screening to before enrollment and during the test
19. Those who drink more than 14 units of alcohol per week within 3 months prior to administration (1 unit of alcohol ≈ 360 mL beer or 45 mL 40% alcohol spirits or 150 mL wine), or those who cannot abstain from alcohol during the study
20. Those who have taken any food or drink that affects absorption, distribution, metabolism, and excretion of the drug within 24 hours before administration, such as food or drink containing caffeine (such as chocolate) and xanthine
21. Those who have consumed pithya , mango, grapefruit, lime, star fruit, or food or beverage prepared therefrom 2 weeks before the first administration
22. Clinically significant clinical laboratory abnormalities or other clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, tumor, pulmonary, immunological, psychiatric or cardiovascular diseases)
23. Those who are positive in urine drug and alcohol test
24. Hepatitis B surface antigen, hepatitis C antibody / hepatitis C core antigen, HIV antigen / antibody, syphilis antibody positive
25. Subjects with other factors not suitable for the trial considered by the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax） | Day 2
Area under the plasma concentration versus time curve (AUC) | Day 2
Peak time in plasma(Tmax) | Day 2
Area under the plasma concentration versus time curve during the dosing interval(AUC0-τ) | Day 9
minimum plasma concentration at steady state(Cmin,ss) | Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China